CLINICAL TRIAL: NCT04122456
Title: Pilot Study on DNA Repair Activity in the Skin of Day and Night Shift Workers
Brief Title: DNA Repair Activity in the Skin of Day and Night Shift Workers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 06753
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Day Shift Work Schedule (Experimental): Day shift worker skin biopsies will be exposed to artificial sunlight (ultraviolet B radiation; UVB) at the laboratory.
  Interventions: Radiation: Ultraviolet B Radiation; Other: No Ultraviolet B Radiation
- Night Shift Work Schedule (Experimental): Night shift worker skin biopsies will be exposed to artificial sunlight (ultraviolet B radiation; UVB) at the laboratory.
  Interventions: Radiation: Ultraviolet B Radiation; Other: No Ultraviolet B Radiation

INTERVENTIONS:
Radiation: Ultraviolet B Radiation — One skin punch biopsy will be taken to the laboratory for exposure to ultraviolet B radiation. After 1-hour incubation, the biopsies will be bisected in half.
Other: No Ultraviolet B Radiation — One skin punch biopsy will be taken to the laboratory and will be kept as a non-irradiated control.

SUMMARY:
The purpose of this study is to test how the skin of night shift workers responds to artificial sunlight (ultraviolet B radiation; UVB) at two different times of the day in comparison to normal day shift workers. After the skin biopsies are obtained, they will be brought to the laboratory to be exposed to UVB radiation and to measure UVB responses.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* Fair skin (Fitzpatrick types I and II)
* Age 18 to 40
* Able to comprehend procedures/risks
* Primarily work and are awake during normal daylight hours (6 am to 6 pm), or primarily work and are awake during night shifts hours (between the hours of 6 pm and 6 am) or may work a mixture of these shifts over the past 3 months. Rotating shifts will be categorized based on the majority of hours worked on average during the last 3 months. Able to fill out a 3-month calendar of work schedule.

Exclusion Criteria:

* Known photosensitivity
* Currently on photosensitizing medications
* Diabetes Mellitus
* On any hormonal agents (e.g., birth control pills)
* History of abnormal scarring
* History of skin infections
* History of skin cancers
* History of sleep disorders such as sleep apnea or insomnia
* Known allergy to lidocaine local anesthetic
* Pregnancy or nursing
* Other serious health issues

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Expression level of the DNA repair factor XPA at two times of the day in the skin of day and night shift workers. | After 1 hour incubation from ultraviolet B radiation exposure.
  Reverse transcription quantitative PCR (RT-qPCR) and immunohistochemistry will be used to measure XPA expression at the mRNA and protein level, respectively, in skin samples obtained at 8 am and 4 pm.
Expression levels of core clock genes at two times of the day in the skin of day and night shift works. | After 1 hour incubation from ultraviolet B radiation exposure.
  Reverse Transcription Quantitative PCR (RT-qPCR) is used to measure the core circadian clock gene expression at the mRNA level in the skin samples obtained at 8 AM and 4 PM.
Activity of the nucleotide excision repair (NER) system at two times of the day in day and night shift workers. | After 1 hour incubation from ultraviolet B radiation exposure.
  A biochemical assay of nucleotide excision repair is used to measure NER in the skin samples obtained at 8 AM and 4 PM.
Activation of DNA damage kinase signaling pathways at two times of the day in the skin of day and night shift workers. | After 1 hour incubation from ultraviolet B radiation exposure.
  Immunohistochemistry is used to measure DNA damage kinase signaling (phosphorylated Chk1 and p53) in the skin samples obtained at 8 AM and 4 PM.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Travers, MD, PhD, Principal Investigator — Wright State University
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT04122456/ICF_000.pdf